CLINICAL TRIAL: NCT03733561
Title: A Randomized, Open-Label, Crossover Study to Evaluate the Pharmacokinetic Profiles of Rotigotine After a Single Dose of LY03003 (28 mg) Versus After a Week of Daily NEUPRO® Transdermal Patch (4 mg Every 24 Hours) in Healthy Volunteers
Brief Title: A Study to Assess Pharmacokinetic Profiles of LY03003 and Neupro
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03003/CT-USA-105
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY03003 (Experimental): LY03003
  Interventions: Drug: LY03003
- Neupro transdermal patch (Active Comparator): Neupro transdermal 4 mg patch
  Interventions: Drug: Neupro 4Mg/24Hr Transdermal Patch

INTERVENTIONS:
Drug: LY03003 — LY03003 (rotigotine extended release microspheres for intramuscular [IM] injection)
  Arms: LY03003
Drug: Neupro 4Mg/24Hr Transdermal Patch — neupro patch
  Arms: Neupro transdermal patch

SUMMARY:
Phase 1, single center study to assess pharmacokinetic profiles of rotigotine after single dose of LY03003 and daily patch application of Neupro in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, subjects must meet all inclusion criteria at screening:

1. Willing and capable of giving informed consent;
2. Between the ages of 18 and 45 years old, inclusive;
3. Healthy, per investigator judgment, based on detailed medical history, clinical laboratory safety tests, vital signs, full physical examination, and ECG;
4. Nonsmoker defined as not having smoked or used any form of tobacco within 6 months before screening;
5. BMI between 18.5 and 30 kg/m2, inclusive, and body weight ≥50 kg at screening;
6. Willing and able to comply with study procedures, adhere to study restriction, and stay at the CRU during in-patient stays required by the protocol;
7. All female subjects (childbearing potential and non-childbearing potential) must have a negative serum pregnancy test result at screening. In addition, female subjects must meet 1 of the following 3 conditions: (i) postmenopausal for at least 12 months without an alternative medical cause, (ii) surgically sterile (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion) based on subject report, or (iii) if of childbearing potential and heterosexually active, practicing or agree to practice a highly effective method of contraception. Highly effective methods of contraception include an intrauterine device (IUD), intrauterine hormone-releasing system (IUS), and contraceptives (oral, skin patches, or implanted or injectable products) using combined or progestogen-only hormonal contraception associated with inhibition of ovulation. A vasectomized male partner is an acceptable contraception method if the vasectomized partner is the sole sexual partner of the female subject and the vasectomized partner has received medical confirmation of surgical success. Highly effective methods of contraception must be used for at least 21 days prior to study drug dosing, throughout the study, and for a minimum of 1 month after the end of the study to minimize the risk of pregnancy.
8. Sexually active, fertile, male patients must be willing to use acceptable contraception methods throughout the study and for at least 1 month after the end of the study if their partners are of childbearing potential.

Exclusion Criteria:

1. History of symptomatic orthostatic hypotension with a decrease of ≥20 mmHg in systolic blood pressure (SBP) or decrease of ≥10 mmHg in diastolic blood pressure (DBP) when changing from a supine to a standing position after having been in the supine position for at least 5 minutes or SBP less than 105 mmHg in a supine position at screening;
2. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, and/or lipid metabolism disorders, and/or drug hypersensitivity;
3. History of epilepsy, seizures as an adult, lifetime history of stroke, or transient ischemic attack (TIA) within 1 year prior to screening;
4. History of sleep attacks or narcolepsy;
5. Known or suspected malignancy within 5 years with the exception of treated and cured basal cell carcinoma (skin), squamous cell carcinoma (skin), or in-situ cervical carcinoma;
6. Positive blood screen for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
7. Positive pregnancy test result or plan to become pregnant if female;
8. Female who is pregnant or breastfeeding or of childbearing potential without adequate contraception (see Inclusion Criterion 7);
9. Hospital admission or major surgery within 30 days prior to screening;
10. Receipt of another investigational product within one month or 5 half-lives of the other investigational product, whichever is longer, before study drug administration in this study.
11. History of prescription drug abuse or any illicit drug use within 6 months prior to screening;
12. History of alcohol abuse according to medical history within 6 months prior to screening;
13. Positive screen for alcohol or drugs of abuse;
14. Unwillingness or inability to comply with food and beverage restrictions during study participation;
15. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
16. Use of prescription or over-the-counter (OTC) medications and/or herbal supplements (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at <3 g/day is permitted until 24 hours prior to dosing);
17. Inability to tolerate study drug in any prior rotigotine or LY03003 trial or intolerance or hypersensitivity to rotigotine or any excipients or diluents (Poly (lactide-co-glycolide) [PLGA], carboxymethylcellulose sodium [SCMC], stearic acid, or mannitol);
18. History of known intolerance/hypersensitivity to antiemetics such as ondansetron, tropisetron, and glycopyrrolate;
19. History of suicide attempt in the past 6 months and/or seen by the investigator as having a significant history of risk of suicide or homicide;
20. Unwillingness of male participants to use appropriate contraceptive measures (see Inclusion Criteria 8) if engaging in sexual intercourse with a female partner of childbearing potential throughout the study and for at least 1 month after the end of the study;
21. Unwillingness to refrain from sexual intercourse with pregnant or lactating women throughout the study and for at least 1 month after the end of the study;
22. Any other clinically relevant hepatic, renal, hematologic, and/or cardiac dysfunction, or other medical condition, or clinically significant laboratory abnormality that would interfere with the subject's safety or study outcome in the judgment of the investigator.
23. A lifetime history of bipolar I disorder, bipolar II disorder, cyclothymia or other specified bipolar and related disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
CMax | 34 days

SECONDARY OUTCOMES:
Adverse Events | 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rivellese, Study Chair — Sponsor GmbH
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No